CLINICAL TRIAL: NCT06580366
Title: Sennosid A+B Versus Sodium Picosulfate/Magnesium Oxide/Citric Acid for Bowel Preparation; A Prospective Randomized Observer-Blinded Study
Brief Title: Comparing Sennosid A+B and Sodium Picosulfate/Magnesium Oxide/Citric Acid for Bowel Preparation
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, İbrahim Durak, Medical Doctor, Hitit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: HititUniversity-2024-43
Record Dates: First submitted 2024-08-27; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Bowel Preparation
Keywords: Bowel preparation; Colonoscopy; sennosid A+B; Sodium Picosulfate
MeSH Terms: interventions — picosulfate sodium

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Sennoside A+B Group" for bowel preparation. (Active Comparator): This study will compare two bowel preparation methods in patients undergoing colonoscopy:
  Sennoside A+B Group
  Intervention: Patients will take Sennoside A+B, a stimulant laxative derived from the senna plant.
  Purpose: To cleanse the colon by increasing bowel movements and reducing water absorption.
  Interventions: Drug: Sennosid A+B
- "PM/Ca Group" for bowel preparation. (Active Comparator): PM/Ca Group (Sodium Picosulfate/Magnesium Oxide/Citric Acid)
  Intervention: Patients will take a combination of sodium picosulfate (a stimulant laxative) and magnesium oxide/citric acid (osmotic agents).
  Purpose: To promote bowel movements by stimulating the bowel and drawing water into the colon.
  Interventions: Drug: Sodium Picosulfate/Magnesium Oxide/Citric Acid

INTERVENTIONS:
Drug: Sennosid A+B — Bowel Preparation
  Arms: "Sennoside A+B Group" for bowel preparation.
Drug: Sodium Picosulfate/Magnesium Oxide/Citric Acid — Bowel Preparation
  Arms: "PM/Ca Group" for bowel preparation.

SUMMARY:
Colonoscopy Preparation: Comparing Sennoside A+B and PM/Ca

Colonoscopy is a test used to examine the inside of the bowel. Proper bowel preparation is crucial because it helps doctors get a clear view during the procedure.

What is Sennoside A+B? Sennoside A+B is a type of laxative made from the senna plant. It works by stimulating the bowel to move and reducing the absorption of water, making it easier to pass stools. Research has shown that high doses of sennoside A+B can be effective for bowel preparation.

Sennoside A+B vs. PEG:

Some studies have found that sennoside A+B is more effective than PEG, another laxative, but can cause more abdominal pain. Other studies have found no significant difference in effectiveness between the two.

What is Picosulfate/Magnesium Oxide/Citric Acid (PM/Ca)? PM/Ca is a combination of sodium picosulfate, magnesium oxide, and citric acid. Sodium picosulfate stimulates bowel movements, while magnesium oxide and citric acid help increase water in the bowel, making it easier to pass stools.

PM/Ca vs. PEG:

Research has shown that PM/Ca is as effective as PEG for bowel preparation. Patients using PM/Ca generally tolerate the preparation process better than those using PEG.

Conclusion:

While PEG is the preferred option according to guidelines, its high cost can make it less accessible in some places. In this study, we aim to compare the effectiveness and patient tolerance of Sennoside A+B and PM/Ca since no direct comparison between these two preparations has been made before.

DETAILED DESCRIPTION:
Colonoscopy is an endoscopic imaging method used to examine the lumen and mucosa of the bowel. It is the gold standard method used for colorectal cancer screening and the detection of most colorectal pathologies. Successful bowel preparation is one of the key factors for a successful colonoscopic examination.

Sennoside A+B is a stimulant laxative derived from the senna plant (Cassia senna). Studies have shown that after senna is ingested, it is activated by the gut flora, directly interacts with the intestinal mucosa, stimulates bowel movements, and inhibits the absorption of electrolytes and water. High doses of senna have been shown to be beneficial as a bowel preparation agent.

There are many studies in the literature comparing senna compounds with polyethylene glycol (PEG) solutions. In a randomized controlled study conducted by Coskun et al. on 474 patients, it was found that bowel cleansing was better with sennoside A+B compared to PEG, but abdominal pain was more common in the senna group. Another randomized controlled study conducted by Shavakhi et al. on 322 patients found no difference in effectiveness between the two agents.

Drugs containing sodium picosulfate-magnesium oxide-citric acid (PM/Ca) are laxative agents recommended for colonoscopy preparation in ESGE and ASGE guidelines. While sodium picosulfate acts as a stimulant laxative, magnesium oxide and citric acid act as osmotic laxatives.

In the SEE CLEAR II randomized controlled trial comparing PM/Ca with PEG, PM/Ca was found to be as effective as PEG. No significant difference was found between the two groups in terms of side effects, but participants using PM/Ca tolerated the bowel preparation procedure much better.

The ASGE and ESGE guidelines primarily recommend PEG solutions for colon preparation. However, due to the lack of reimbursement by the Social Security Institution (SGK) in our country and the resulting cost, access to PEG treatment is difficult for patients. For these reasons, other treatments recommended in the available guidelines are used more frequently in our country.

Although there are many studies in the literature comparing PM/Ca and sennoside A+B preparations with PEG and other preparations in terms of efficacy for bowel preparation, no study has directly compared PM/Ca with sennoside A+B to date. We aimed to compare the efficacy and patient tolerance of these two commonly used preparations in our country.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-80 years scheduled for elective outpatient colonoscopy.
* Ability to provide informed consent.

Exclusion Criteria:

* History of intra-abdominal surgery.
* Chronic kidney failure.
* Congestive heart failure.
* Chronic liver failure.
* Inflammatory bowel disease.
* Electrolyte imbalance.
* Hospitalized patients.
* Patients unable to use the bowel preparation treatment
* Known allergy or hypersensitivity to Sennoside A+B or PM/Ca components
* Known gastrointestinal motility disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-08-22 (Estimated); Primary Completion 2024-12-22 (Estimated); Study Completion 2025-03-22 (Estimated)

PRIMARY OUTCOMES:
Sennosid A+B versus Sodium Picosulfate/Magnesium Oxide/Citric Acid for Bowel Preparation: A Prospective Randomized Observer-Blinded Study | 4 months
  Effectiveness of bowel preparation using the Boston Bowel Preparation Scale (BBPS).
  The BBPS is a standardized 9-point assessment scale for the colon. The structure of the colon is divided into its three segments: right colon, transverse colon, and left colon. Each segment is classified from 0 to 3 depending on the degree of soiling. The sum total of the three segments represents the degree of soiling, so that a total ≤ 5 points shows poor bowel preparation, while 6-7 shows good bowel preparation, and ≥ 8 very good bowel preparation. The investigators will consider patients with a score of 6 or higher as successful.

CONTACTS AND LOCATIONS:
Overall Officials: İbrahim Durak, Study Chair — Hitit University
Locations (1):
- Hitit University Erol Olcok Training and Research Hospital, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Park S, Lim YJ. Adjuncts to colonic cleansing before colonoscopy. World J Gastroenterol. 2014 Mar 21;20(11):2735-40. doi: 10.3748/wjg.v20.i11.2735. PMID 24659864
- [Background] Coskun Y, Yuksel I. Polyethylene glycol versus split high-dose senna for bowel preparation: A comparative prospective randomized study. J Gastroenterol Hepatol. 2020 Nov;35(11):1923-1929. doi: 10.1111/jgh.15101. Epub 2020 Jun 8. PMID 32424868
- [Background] Shavakhi A, Kianinia M, Torabi G, Nemati A, Saeidian B, Hoseinzadeh M, Madjlesi F, Navaei P, Rashidinejad F, Minakari M. High dose Senna or Poly Ethylene Glycol (PEG) for elective colonoscopy preparation: a prospective randomized investigator-blinded clinical trial. J Res Med Sci. 2011 Feb;16(2):149-55. PMID 22091224
- [Background] Katz PO, Rex DK, Epstein M, Grandhi NK, Vanner S, Hookey LC, Alderfer V, Joseph RE. A dual-action, low-volume bowel cleanser administered the day before colonoscopy: results from the SEE CLEAR II study. Am J Gastroenterol. 2013 Mar;108(3):401-9. doi: 10.1038/ajg.2012.441. Epub 2013 Jan 15. PMID 23318484
- [Background] Hassan C, East J, Radaelli F, Spada C, Benamouzig R, Bisschops R, Bretthauer M, Dekker E, Dinis-Ribeiro M, Ferlitsch M, Fuccio L, Awadie H, Gralnek I, Jover R, Kaminski MF, Pellise M, Triantafyllou K, Vanella G, Mangas-Sanjuan C, Frazzoni L, Van Hooft JE, Dumonceau JM. Bowel preparation for colonoscopy: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Update 2019. Endoscopy. 2019 Aug;51(8):775-794. doi: 10.1055/a-0959-0505. Epub 2019 Jul 11. PMID 31295746